CLINICAL TRIAL: NCT03777969
Title: Precise Prediction System for Clinical Endpoint Events of Chronic Hepatitis B Patients in the Ear of Antiviral Therapy
Brief Title: Prediction System of Clinical Endpoint Events for Chronic Hepatitis B Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Ruijin Hospital (Other); ShuGuang Hospital (Other); Beijing Ditan Hospital (Other); Hangzhou Choutu Technology Co.,Ltd. (Unknown); Wuxi Hisky Medical Technologies Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Hong You, Vice President of Beijing Friendship Hospital, Beijing Friendship Hospital
Other Study IDs: 2018ZX10302204-001
Record Dates: First submitted 2018-10-27; First posted 2018-12-19 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic Hepatitis B; Liver fibrosis/cirrhosis; HBV-related endpoint events; Precise prediction model
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Liver biopsy and peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 2000 chronic hepatitis B (CHB) patients with liver biopsy performed at least 1 year after antiviral therapy are enrolled. All the patients will receive original antiviral treatment for the following 10 years. Patients will be assessed at baseline and at every six months for blood count, liver function test, alpha fetoprotein (AFP), prothrombin time, liver ultrasonography, liver stiffness measurement (LSM), Hepatitis B virus (HBV) DNA and HBV serological markers. HBV-related endpoint events, including cirrhosis decompensations (ascites, esophageal variceal bleeding and hepatic encephalopathy), hepatocellular carcinoma (HCC), liver transplantation and liver-related death, will be collected during follow-up.

DETAILED DESCRIPTION:
No.

ELIGIBILITY:
Group 1: Patients with history of HBV-related clinical endpoint events

Inclusion Criteria:

* No age limit;
* Male or female;
* Patients with liver biopsy performed at least 1 year after antiviral therapy; patients with history of clinical endpoint events (decompensated cirrhosis, hepatocellular carcinoma, liver transplantation or liver-related death) after liver biopsy;
* Patients with liver biopsy or liver stiffness or aspartate aminotransferase (AST)-to-platelet (PLT) ratio index (APRI) before antiviral treatment.

Exclusion Criteria:

* Patients with decompensated cirrhosis (including ascites, hepatic encephalopathy, esophageal varices bleeding, hepatorenal syndrome, spontaneous bacterial peritonitis, or other complications of decompensated cirrhosis), hepatocellular carcinoma, or liver transplantation before liver biopsy;
* Patients with hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection, alcoholic liver disease, autoimmune liver disease, genetic liver disease, drug-induced liver injury, or other chronic liver diseases;
* Patients with malignant lesion on liver image;
* Patients with other uncured malignant tumors;
* Patients with severe heart, lung, kidney, brain, blood, neuropsychiatric or other organs diseases;
* Pregnant or lactating women;
* Patients with any other reasons not suitable for the study.

Group 2: Patients without history of clinical endpoint events

Inclusion Criteria:

* No age limit;
* Male or female;
* Patients with liver biopsy performed at least 1 year after antiviral therapy; or chronic hepatitis B (CHB) patients with antiviral therapy at least 1 year content to be performed liver biopsy at enrollment;
* Patients with liver biopsy or liver stiffness or APRI before antiviral treatment;
* Agree to be followed up regularly;
* Signature of informed consent.

Exclusion Criteria:

* Patients with decompensated cirrhosis (including ascites, hepatic encephalopathy, esophageal varices bleeding, hepatorenal syndrome, spontaneous bacterial peritonitis, or other complications of decompensated cirrhosis), hepatocellular carcinoma, or liver transplantation;
* Patients with HCV or HIV infection, alcoholic liver disease, autoimmune liver disease, genetic liver disease, drug-induced liver injury, or other chronic liver diseases;
* Patients with malignant lesion on liver image;
* Patients with other uncured malignant tumors, exclude who were cured;
* Patients with severe heart, lung, kidney, brain, blood, neuropsychiatric or other organs diseases;
* Pregnant or lactating women;
* Patients with any other reasons not suitable for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CHB patients with liver biopsy performed at least 1 year after antiviral therapy; or CHB patients with antiviral therapy for at least 1 year content to be performed liver biopsy at enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
HBV-related clinical endpoint events, including liver decompensations (ascites, esophageal variceal bleeding and hepatic encephalopathy), HCC, liver transplantation and liver-related death | 1 to 10 years
  Incidence of HBV-related clinical endpoint events during follow-ups

SECONDARY OUTCOMES:
Predicted probability of HBV-related clinical endpoint events | 1 to 10 years
  The predicted probability is measured by histological prediction model or non-invasive prediction model
Predicted probability of HBV-induced fibrosis/cirrhosis regression | 1 to 10 years
  The predicted probability is measured by histological prediction model or non-invasive prediction model
Percentage of HBV-induced liver fibrosis/cirrhosis regression | 1 to 10 years
  Liver fibrosis regression was defined as decrease >= 1 point by Ishak fibrosis scoring system (range from 0 to 6, higher values represent a worse outcome) or Predominantly Regressive in P-I-R ( predominantly progressive, indeterminate and predominately regressive) score

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (7):
- China (7):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Wuxi Hisky Medical Technologies Co., Ltd., Wuxi, Jiangsu
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shuguang Hospital affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Hangzhou Choutu Technology Co.,Ltd., Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Chen W, Chen S, Wu X, Zhang X, Zhang L, Zhao H, Xu M, Chen Y, Piao H, Li P, Li L, Jiang W, Li X, Xing H, Liu X, Zhang Y, Wang B, Zhou J, Meng T, Zhao X, Shao C, Kong Y, Zhao X, Ou X, Liu C, Jia J, You H. Regression of Liver Fibrosis in Patients on Hepatitis B Therapy Is Associated With Decreased Liver-Related Events. Clin Gastroenterol Hepatol. 2024 Mar;22(3):591-601.e3. doi: 10.1016/j.cgh.2023.11.017. Epub 2023 Nov 30. PMID 38040276